CLINICAL TRIAL: NCT07391293
Title: Genetic Aortic Diseases and Cardiovascular Complications. An Observational Survey of Risk Factors.
Acronym: PROM-1
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alessandro Pini, MD, IRCCS Policlinico S. Donato
Other Study IDs: PROM-1
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Thoracic Aortic Aneurysm (TAA)
Keywords: risk stratification; quality of life; rare disease; survey
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Rare Diseases | interventions — Quality of Life; Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAA: subjects with TAA aged between 14 and 60 years
  Interventions: Other: Journey to diagnosis; Other: Quality of life, functional health and well-being; Other: Awareness and self-esteem, acceptance of the condition; Other: psychological and physical well-being

INTERVENTIONS:
Other: Journey to diagnosis — Questions relating to the course and experience/history of the disease from the onset of symptoms to confirmation of diagnosis; accessibility to referral facilities for treatment and follow-up.
Other: Quality of life, functional health and well-being — Qestionnaires
Other: Awareness and self-esteem, acceptance of the condition — questionnaire related to the quality of life and self-care
Other: psychological and physical well-being — questionnaire to describe psychological and physical well-being.

SUMMARY:
The aim of this observational study is to define the behavioural and cardiovascular risk factor profiles of patients with genetic aortopathies. The main questions it aims to answer are:

* How do the interconnections between lifestyle, stress, psychological condition, perception of illness, and state of health influence each other in this population?
* Beyond traditional risk factors, additional emerging factors should be considered, including pregnancy-related complications, sedentary lifestyle, early menopause and depression. The interplay between eating disorders, lifestyle factors and autoimmune or inflammatory bowel diseases remains poorly understood.

DETAILED DESCRIPTION:
Thoracic aortic aneurysms (TAA) present peculiar symptoms as well as high mortality due to complications related to dilatation and dissection of the ascending aorta and great arteries. The presence or absence of extra-aortic features determines whether TAADs are syndromic, associated with diseases affecting other systems and organs, or non-syndromic, with manifestations limited to the aorta. Life expectancy of patients withTAA has improved markedly in the last decades, but still remains lower than that of the general population.

ELIGIBILITY:
Inclusion Criteria:

* signed onformed consent
* Ability to speak, read and write in Italian

Exclusion Criteria:

-

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with TAA either syndromic or non-syndromic followed at the Cardiovascular Genetic Centre, IRCCS Policlinico San Donato
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Journey to diagnosis | 15 months
  The mean, median, standard deviation and interquartile range will be used for continuous variables, whereas frequency and percentage will be applied for nominal and categorical variables. The Shapiro-Wilks test will be used to assess the Gaussian distributions.
Quality of life, functional health and well-being | 15 months
  The mean, median, standard deviation and interquartile range will be used for continuous variables, whereas frequency and percentage will be applied for nominal and categorical variables. The Shapiro-Wilks test will be used to assess the Gaussian distributions.
Awareness and self-esteem, acceptance of the condition | 15 months
  The mean, median, standard deviation and interquartile range will be used for continuous variables, whereas frequency and percentage will be applied for nominal and categorical variables. The Shapiro-Wilks test will be used to assess the Gaussian distributions.
psychological and physical well-being | 15 months
  The mean, median, standard deviation and interquartile range will be used for continuous variables, whereas frequency and percentage will be applied for nominal and categorical variables. The Shapiro-Wilks test will be used to assess the Gaussian distributions.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Policlinico San Donato, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
PD will not or might not be shared according to the preliminary results

REFERENCES:
- [Background] Saeyeldin, Ayman A., Camilo A. Velasquez, Syed Usman B. Mahmood, Adam J. Brownstein, Mohammad A. Zafar, Bulat A. Ziganshin, e John A. Elefteriades. 2019. "Thoracic aortic aneurysm: unlocking the "silent killer" secrets". General Thoracic and Cardiovascular Surgery 67(1):1-11.
- [Background] Udugampolage, Nathasha, Rosario Caruso, Mariangela Panetta, Edward Callus, Federica Dellafiore, Arianna Magon, Susan Marelli, e Alessandro Pini. 2021. "Is SF-12 a valid and reliable measurement of health-related quality of life among adults with Marfan syndrome? A confirmatory study". PLoS ONE 16(6 June):e0252864. doi: 10.1371/journal.pone.0252864.